CLINICAL TRIAL: NCT01012154
Title: In Vivo Confocal Microscopy Tumor Atlas Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carl Zeiss Surgical GmbH (Industry)
Responsible Party: Dr. Gerhard Gaida / Clinical Affairs, Carl Zeiss Surgical GmbH
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 002874
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2009-11-11 (Estimated); Status verified 2009-11

CONDITIONS: Brain Neoplasms
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients (Experimental)
  Interventions: Device: Endomicroscope

INTERVENTIONS:
Device: Endomicroscope — Endomicroscopic images and biopsies are taken at several positions on the tumor.

SUMMARY:
This study aims to create an atlas based on the preliminary experience of the first feasibility study in neurosurgery. Hypothesis: That a confocal endomicroscope can be used during neurosurgery to provide in vivo histology that enables documentation of neurological pathology across a range of tumor ypes and grades, suitable for comparison with traditional histopathology from site-matched biopsies.

DETAILED DESCRIPTION:
Confocal endomicroscopy is a medical imaging modality that allows real-time microscopy to be performed on living tissue in vivo. The procedure involves a small endoscope which is placed gently into contact with the tissue, providing significant in vivo magnification on a scale similar to that obtained by the pathology laboratory microscope. It is already in clinical use in the field of gastroenterological endoscopy, and investigational use in laparoscopy, dermatology and gynecology. Further, in recent pilot studies endomicroscopy has also been shown to be feasible in bronchoscopy, robot assisted prostatectomy and neurosurgery.The study will use both endomicroscopy and biopsy to document the histological appearance of a range of neurological tumour types and grades.

In subsequent analysis, the confocal image data and corresponding histology data and images will be used to document reliably observable features in the confocal images that are relevant to histopathology interpretation. Relevant images will be selected and discussed by comparison to frozen or permanent section histology for compilation into an atlas documenting comparison for the tumors seen in the study.

ELIGIBILITY:
Inclusion Criteria:

* All patients with neurological pathology requiring surgery in which tumour resection might be evaluated by using biopsy

Exclusion Criteria:

* History of allergy to fluorescein
* Patients on beta-blockers or ACE inhibitors
* Pregnant women
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Generation of an atlas documenting the comparative features of in vivo microscopy versus traditional histopathology of site-matched biopsies across a range of tumor types and grades. | During surgery

SECONDARY OUTCOMES:
Test the ability of an expert neuropathologist to predict the outcome of biopsies based on the confocal images collected in vivo. | One week
Capture usability and workflow aspects for the confocal device. | During surgery

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nakaji, MD, Principal Investigator — Barrow Neurological Institute, St. Joseph's Hospital and Medical Center
Locations (1):
- Barrow Neurological Institute, St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States